CLINICAL TRIAL: NCT05088044
Title: A Quasi Experimental Study to Assess the Impact of Implementing Modified Early Warning Score in Terms of Competency and Self-efficacy of Nurses at ILBS, Delhi
Brief Title: A Study to Assess the Impact of Implementing Modified Early Warning Score in Terms of Competency and Self-efficacy of Nurses at ILBS, Delhi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ILBS-Liver Disease-01
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2021-10

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: one group pre-test post-test design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- staff nurses (Experimental): firstly pre-test would conducted for the group then after 7 days post-test would be conducted for the same group intervention which will be given: training on modified early warning score to staff nurses and marking of physiological parameters on MEWS chart
  Interventions: Other: training porogram

INTERVENTIONS:
Other: training porogram — training on modified early warning signs will be given to staff nurses and they will be asked to mark physiological parameters on MEWS chart and identify detrioration

SUMMARY:
In this study nurses will be taught regarding Modified Early Warning Score and how to mark the involved physiological parameters in the MEWS chart and then scoring will be given i.e MEWS score and according to the score intervention would be taken by nurses by communicating with other health team members. this scoring will allow nurses to assess early deterioration and early ICU admission and at last nurses will be asked regarding the barriers or facilitators they faced while performing MEWS score.

ELIGIBILITY:
Inclusion Criteria:

* registered nurses working in general, semi-private and private ward nurses willing to participate

Exclusion Criteria:

* registered nurses who will not be present at the time of data collection. pull out staffs.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
to assess the impact of MEWS on competency and self-efficacy of nurses before and after implementing MEWS | 7 days
  pre-test would be taken to assess previous level and post-test to measure the change in competency

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No